CLINICAL TRIAL: NCT01447576
Title: A Phase 2, Multicenter, Open-label Study to Assess the Safety and Tolerability of Oral OPC-34712 as Adjunctive Therapy in Adult Patients With Major Depressive Disorder
Brief Title: Study of Safety & Tolerability of OPC-34712 as Adjunctive Therapy in Treatment of Adult Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 331-08-212
Record Dates: First submitted 2011-09-29; First posted 2011-10-06 (Estimated); Results first posted 2015-11-06 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-10

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OPC-34712 + ADT (Experimental): Experimental: OPC-34712, Oral Tablets, 0.25 - 3 mg; Antidepressant drug treatment
  Interventions: Drug: ADT; Drug: OPC-34712

INTERVENTIONS:
Drug: ADT — Once daily dosing during the duration of the study.
  Other Names: Anti-depressant Drug Therapy
Drug: OPC-34712 — OPC-34712, Oral Tablets, 0.25 - 3 mg

SUMMARY:
The purpose of this study is to assess the long-term safety, tolerability and efficacy of oral OPC-34712 as adjunctive therapy in the treatment of adult patients with Major Depressive Disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 18 and 65 years of age, with a diagnosis of a single or recurrent, non-psychotic episode of major depressive disorder, as defined by DSM-IV-TR criteria and confirmed by the Mini International Neuropsychiatric Interview (M.I.N.I.) which is equal to or greater than 8 weeks in duration.
* Subjects must currently be taking allowable antidepressant therapy at an adequate dose for a minimum of six weeks by the end of the screening period (ie at the time of the Baseline visit).
* Subjects must report a history for the current depressive episode of an inadequate response to at least one and no more than four adequate antidepressant treatments.

Exclusion Criteria:

* Females who are breast-feeding and/or who have a positive pregnancy test result prior to receiving study drug.
* Subjects who report an inadequate response to more than three adequate trials of antidepressant treatments during current depressive episode at a therapeutic dose for an adequate duration.
* Subjects with a current Axis I (DSM-IV-TR) diagnosis of: Delirium, dementia,amnestic or other cognitive disorder Schizophrenia, schizoaffective disorder, or other psychotic disorder Bipolar I or II disorder, eating disorder (including anorexia nervosa or bulimia), obsessive compulsive disorder, panic disorder, post-traumatic stress disorder.
* Subjects with a clinically significant current Axis II (DSM-IV-TR) diagnosis of borderline, antisocial, paranoid, schizoid, schizotypal or histrionic personality disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1036 (Actual)
Dates: Start 2009-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- United States (32):
  - Pacific Clinical Research Medical Group, Arcadia, California
  - Artemis Institute for Clinical Research, San Diego, California
  - California Neuroscience Research Medical Group, Inc., Sherman Oaks, California
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - Clinical Neuroscience Solutions, Jacksonville, Florida
  - Florida Clinical Research Center, Maitland, Florida
  - Clinical Neurosciences Solutions, Orlando, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Carman Research, Smyrna, Georgia
  - Goldpoint Clinical Research, LLC, Indianapolis, Indiana
  - Pharmasite Research, Baltimore, Maryland
  - Clinical Insights, Glen Burnie, Maryland
  - Rochester Center for Behavioral Medicine, Rochester Hills, Michigan
  - Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Brooklyn Medical Institute, Brooklyn, New York
  - Medical & Behavioral Health Research, New York, New York
  - The Medical Research Network, LLC, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Midwest Clinical Research Center, Dayton, Ohio
  - Oregon Center for Clinical Investigations, Inc., Portland, Oregon
  - Oregon Center for Clinical Investigations, Salem, Oregon
  - Carolina Clinical Research Services, Columbia, South Carolina
  - FutureSearch Trials of Dallas, Dallas, Texas
  - Bayou City Research, Ltd., Houston, Texas
  - Radiant Research, Murray, Utah
  - Psychiatric Alliance of the Blue Ridge, Charlottesville, Virginia
  - Neuroscience, Inc., Herndon, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Summit Research Network, Seattle, Washington
  - Northbrooke Research Center, Brown Deer, Wisconsin
  - Dean Foundation, Middleton, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1036 participants entered trial, including 792 who had rolled over from previous studies and 244 de novo participants. Of the 792 rollovers, 337 were 6-week enrollers and the 52-week enrollers consisted of 699 enrolled participants (455 rollover and 244 de novo). This was a single arm study and all participants received the same treatment.
Pre-assignment Details: Eligible participants received daily treatment with open-label brexpiprazole (0.25 up to 3.0 milligrams (mg)/day) and commercially marketed ADT.
Groups:
- Brexpiprazole +ADT: All participants received brexpiprazole 0.25 to 3.0 mg/day plus ADT.
Period: Overall Study
Arm/Group | Brexpiprazole +ADT
Started | 1036
Completed | 560
Not Completed | 476
Not completed — Lost to Follow-up | 52
Not completed — Adverse Event | 127
Not completed — Participant met withdrawal criteria | 40
Not completed — Withdrawal by Subject | 100
Not completed — Protocol deviation | 83
Not completed — Lack of Efficacy | 68
Not completed — Physician Decision | 6

BASELINE CHARACTERISTICS:
Groups:
- Brexpiprazole+ADT: All participants received brexpiprazole 0.25 to 3.0 mg/day plus ADT.
Arm/Group | Brexpiprazole+ADT
Number analyzed (Participants) | 1036
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.0 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 702
  Male | 334

OUTCOME MEASURES:

1. Primary Outcome: Participants With Adverse Events (AEs).
Description: An AE was defined as any new medical problem, or exacerbation of an existing problem, experienced by a participant while enrolled in the trial, whether or not it was considered drug-related by the physician. The severity was assessed as mild, moderate, or severe. A treament-emergent AE (TEAE) was defined as any AE that started after start of open-label brexpiprazole; or if the event was continuous from baseline and was worsening, serious, study drug-related, or resulted in death, discontinuation, interruption, or reduction of study drug.
Time Frame: After the Informed Consent Form (ICF) was signed, through Follow up 30 (+2) days after last visit
Population: The primary safety dataset included all participants exposed to at least 1 dose of brexpiprazole.
Measure: Number; unit: Participants
Arm/Group | Brexpiprazole+ADT
Number analyzed (Participants) | 1034
Participants
  Participants with TEAEs | 851
  Participants with serious TEAEs | 30

2. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity of Illness (CGI-S) Scale Score.
Description: The CGI-S is a 7-point scale from 1 through 7. The items on CGI-S scale are: 0 = not assessed, 1 = normal, not at all ill, 2 = borderline mentally ill, 3 = mildly ill, 4 = moderately ill, 5 = markedly ill, 6 = severely ill, 7 = among the most extremely ill participants. The score 0 (= not assessed) was set to missing.
Time Frame: Week 1, 2, 4, 6, 8, 14, 20, 26, 32, 38, 44, 52 and 52 (last-observation-carried-forward [LOCF])
Population: Efficacy dataset had participants who received at least 1 dose of brexpiprazole and had a baseline and at least 1 postbaseline efficacy evaluation for CGI-S. LOCF dataset included data recorded at a given visit in treatment phase or, if no observation was recorded at that visit, data carried forward from the previous visit in the Treatment Phase.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Brexpiprazole+ADT
Number analyzed (Participants) | 1032
Units on a scale
  Week 1 | -0.09 (0.60)
  Week 2 | -0.35 (0.82)
  Week 4 | -0.63 (0.96)
  Week 6 | -0.79 (1.03)
  Week 8 | -0.92 (1.12)
  Week 14 | -0.93 (1.14)
  Week 20 | -1.08 (1.17)
  Week 26 | -1.13 (1.24)
  Week 32 | -1.24 (1.24)
  Week 38 | -1.37 (1.28)
  Week 44 | -1.46 (1.27)
  Week 52 | -1.52 (1.34)
  Week 52-LOCF | -0.81 (1.24)

3. Secondary Outcome: Mean Clinical Global Impression - Improvement (CGI-I) Scale Score.
Description: The items on CGI-I scale are 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, 7 = very much worse. The score of 0 (= not assessed) was set to missing. The CGI-I is therefore a 7-point scale from 1 through 7. CGI improvement was compared to the participants condition at Baseline.
Time Frame: Week 1, 2, 4, 6, 8, 14, 20, 26, 32, 38, 44, 52 and 52 (LOCF)
Population: Efficacy dataset had participants who received at least 1 dose of brexpiprazole and had a baseline and atleast 1 postbaseline efficacy evaluation for CGI-S. LOCF dataset included data recorded at a given visit in treatment phase or, if no observation was recorded at that visit, data carried forward from the previous visit in the Treatment Phase.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Brexpiprazole+ADT
Number analyzed (Participants) | 1023
Units on a scale
  Week 1 | 3.38 (0.94)
  Week 2 | 3.04 (1.06)
  Week 4 | 2.67 (1.09)
  Week 6 | 2.46 (1.10)
  Week 8 | 2.36 (1.10)
  Week 14 | 2.36 (1.23)
  Week 20 | 2.22 (1.17)
  Week 26 | 2.16 (1.12)
  Week 32 | 2.08 (1.13)
  Week 38 | 1.97 (1.11)
  Week 44 | 1.91 (1.14)
  Week 52 | 1.92 (1.15)
  Week 52-LOCF | 2.57 (1.31)

ADVERSE EVENTS:
Time Frame: After the ICF was signed, through the treatment period and through Follow-up (telephone contact or in-clinic visit) 30 (+ 2) days after the last visit.
Description: The safety sample consisted of participants who received at least 1 dose of brexpiprazole. Serious adverse event data were available for 697 participants (52 Week enrollers). Non-serious AE data were available for 1034 participants.
Groups:
- Brexpiprazole+ADT: Participants received brexpiprazole 0.25 to 3.0mg/day plus ADT.
Arm/Group | Brexpiprazole+ADT
Serious Adverse Events (participants affected / at risk) | 29/697
Other Adverse Events (participants affected / at risk) | 684/1034
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole+ADT (N=697)
Pancreatitis (Gastrointestinal disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Pneumonia (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Intentional overdose (Injury, poisoning and procedural complications) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Convulsion (Nervous system disorders) | 1
Cranial nerve paralysis (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Anxiety (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 3
Depression suicidal (Psychiatric disorders) | 1
Depressive symptom (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 3
Suicide attempt (Psychiatric disorders) | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole+ADT (N=1034)
Fatigue (General disorders) | 95
Upper respiratory tract infection (Infections and infestations) | 67
Weight increased (Investigations) | 217
Increased appetite (Metabolism and nutrition disorders) | 87
Akathisia (Nervous system disorders) | 102
Dizziness (Nervous system disorders) | 60
Headache (Nervous system disorders) | 87
Sedation (Nervous system disorders) | 54
Somnolence (Nervous system disorders) | 94
Tremor (Nervous system disorders) | 42
Anxiety (Psychiatric disorders) | 67
Insomnia (Psychiatric disorders) | 91
Restlessness (Psychiatric disorders) | 59
Constipation (Gastrointestinal disorders) | 41
Diarrhoea (Gastrointestinal disorders) | 42
Dry mouth (Gastrointestinal disorders) | 40
Nausea (Gastrointestinal disorders) | 50
Nasopharyngitis (Infections and infestations) | 47
Back pain (Musculoskeletal and connective tissue disorders) | 33
Abnormal dreams (Psychiatric disorders) | 41
Middle insomnia (Psychiatric disorders) | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No